CLINICAL TRIAL: NCT07154771
Title: Development and Usability Evaluation of an Arm Circumference Measurement Tool For Patients Undergoing Breast Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Rumeysa Ozcelik, Research Assistant, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2025-347
Record Dates: First submitted 2025-07-21; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Breast Surgery; Breast Cancer; Lymphedema
Keywords: breast cancer; mastectomy; nursing; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two phases: the first phase involves the development of the arm circumference measurement device, and the second phase consists of a two-group crossover randomized controlled trial to evaluate the usability of the developed device.
  Within this scope, the intra-observer and inter-observer reliability of the traditional tape measure and the newly developed arm circumference measurement device for measuring upper extremity circumference will be compared. In the crossover design, nurses and patients will be randomly assigned to study groups where both measurement methods will be applied in a predetermined order. There are a total of four study groups for nurses and patients, based on intervention-control and control-intervention sequences.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participants (patients and nurses) and the statistician conducting the data analyses are blinded to the group assignments of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- İntervention-control group (Patient) (Other): The intervention-control group will first perform circumference measurements using the arm circumference measurement device, followed by measurements with the tape measure. The measurement values obtained by the patients will be recorded in the Anthropometric Measurement and Time Tracking Form. The researcher will use a stopwatch to record the duration of the measurements, which will also be documented in the form.
  Interventions: Other: First with the arm circumference measurement tool, then with the traditional tape measure
- Control-Intervention Group (Patients) (Other): The control-intervention group will first perform circumference measurements using the tape measure, followed by measurements with the arm circumference measurement device. The measurement values obtained by the patients will be recorded in the Anthropometric Measurement and Time Tracking Form. The researcher will use a stopwatch to record the duration of the measurements, which will also be documented in the form.
  At the end of the procedure, all patients will complete the Visual Analog Scale (VAS), Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST), and Patient Interview Form.
  Interventions: Other: First with the traditional tape measure , then with the arm circumference measurement tool
- Intervention-Control Group (Nurses) (Other): The intervention-control group will first perform circumference measurements using the arm circumference measurement device, followed by measurements with the tape measure. Nurses will record their measurement values in the Anthropometric Measurement and Time Tracking Form. The researcher will use a stopwatch to record the duration, which will also be noted in the form.
  Interventions: Other: First with the arm circumference measurement tool, then with the traditional tape measure
- Control-Intervention Group (Nurses) (Other): The control-intervention group will first perform circumference measurements using the tape measure, followed by measurements with the arm circumference measurement device. Nurses will record their measurement values in the Anthropometric Measurement and Time Tracking Form. The researcher will use a stopwatch to record the duration, which will also be noted in the form.
  At the end of the procedure, all nurses will complete the Visual Analog Scale (VAS), Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST), and Nurse Interview Form.
  Interventions: Other: First with the traditional tape measure , then with the arm circumference measurement tool

INTERVENTIONS:
Other: First with the arm circumference measurement tool, then with the traditional tape measure — Patients and nurses in this group will measure both arms (at four different anatomical reference points) first using the newly developed arm circumference measurement device, followed by the traditional tape measure.
  Arms: Intervention-Control Group (Nurses); İntervention-control group (Patient)
Other: First with the traditional tape measure , then with the arm circumference measurement tool — Patients and nurses in this group will measure both arms (at four different anatomical reference points) first using the traditional tape measure, and then using the newly developed arm circumference measurement device.
  Arms: Control-Intervention Group (Nurses); Control-Intervention Group (Patients)

SUMMARY:
The aim of this study is to develop an arm circumference measurement device that can be used by both patients and nurses in the follow-up of upper extremity lymphedema, which may occur as a result of breast cancer surgery, and to evaluate its usability. This study also seeks to determine whether the developed device can offer a more accurate, faster, and more practical alternative compared to traditional tape measurements. The main questions it aims to answer are:

Is there a significant difference in intra-observer reliability between the measurements taken by nurses and patients using the arm circumference measurement device and those taken using a traditional tape measure?

Is there a significant difference in inter-observer reliability between the measurements taken by nurses and patients using the arm circumference measurement device and those taken using a traditional tape measure?

Is there a significant difference in the measurement results obtained by nurses and patients when using the arm circumference measurement device compared to a traditional tape measure?

Do nurses and patients experience a difference in the duration of arm circumference measurements when using the measurement device versus a traditional tape measure?

Is there a difference in the satisfaction levels of nurses and patients regarding arm circumference measurements performed with the measurement device versus a traditional tape measure? This study will be conducted in two phases: the first phase involves the development of the arm circumference measurement tool, and the second phase involves the evaluation of its usability through a double-blind, two-group, crossover randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

Nurses:

-Currently working in General Surgery or Surgical Oncology clinics

Patients:

* Aged 18 years or older
* Newly diagnosed with breast cancer confirmed by histopathology
* Planned to undergo radical mastectomy, modified radical mastectomy, or breast-conserving surgery
* Scheduled for axillary lymph node dissection (at least two lymph nodes to be dissected)
* Able to understand information related to circumference measurement and perform the required skills

Exclusion Criteria:

Patients:

* Patients who have undergone bilateral lymph node dissection
* Patients with a prior diagnosis and treatment for breast cancer (surgery, chemotherapy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the study focuses on breast cancer, which is the most common cancer type among women worldwide, patient participants are required to be female. However, nurse participants can be of any gender.
Enrollment: 35 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Intra-rater Reliability | Preoperative period (Same day, within 30 minutes between repeated measurements.) The same rater (nurse/patient/researcher) performs repeated measurements on the same arm with both methods within a short interval to assess consistency.
  The consistency of repeated measurements performed by the same individual (nurse, patient, or researcher) using different methods (tape measure and the newly developed arm circumference measurement device).
  Evaluated separately for the right and left arms.
  Comparisons will be made between the two measurement methods.
Inter-rater Reliability | Preoperative period (Same day, sequential measurements within 1 hour by different raters.) Measurements by different raters (nurse, patient, researcher) are conducted on the same day in a fixed sequence.
  The agreement between different raters (nurse-patient, nurse-researcher, patient-researcher) using the same method (either tape measure or the new measurement device).
  Evaluated for both arms and both measurement tools.
  Inter-rater agreement will be assessed across all rater combinations.

SECONDARY OUTCOMES:
Measurement Duration | Preoperative period (all measurements for both arms; each method's duration recorded separately and immediately)
  For each participant (both nurse and patient), the duration of each measurement-performed on both the right and left arms using both the tape measure and the arm circumference measurement device-will be recorded using a stopwatch. These same-day measurements will be used to compare the time efficiency and practicality of the two methods.
  Comparison will be made between the two methods in terms of time efficiency and practicality.
User Satisfaction - Visual Analog Scale (VAS) | Preoperative period (each participant completes both measurement methods; immediately after finishing all measurements for both arms, the participant completes the same-day questionnaire without delay)
  Nurses' and patients' satisfaction with each measurement method will be assessed using a Visual Analog Scale ranging from 0 (not satisfied at all) to 10 (completely satisfied).
  Differences in satisfaction between methods and arms will be analyzed.
User Satisfaction - Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) | Preoperative period (questionnaire completed immediately after all measurements on both arms using both methods)
  Satisfaction with the new measurement device will be evaluated using the standardized QUEST 2.0 questionnaire, which assesses satisfaction with assistive devices and related services.
  Higher scores indicate higher levels of satisfaction.
  Administered to both nurses and patients.
Open-ended Feedback (Interview Forms) | Preoperative period (open-ended feedback collected immediately after completing both measurement methods and satisfaction scales during the same session) Türkçe:
  Qualitative data will be collected through structured interview forms to explore the experiences, perceptions, and suggestions of nurses and patients regarding the use of the new arm circumference measurement device.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice AYHAN, Professor, Study Director — SBUniversite
Locations (1):
- Gülhane Training and Research Hospital, University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not intend to share individual participant data (IPD).

REFERENCES:
- [Background] Zou L, Liu FH, Shen PP, Hu Y, Liu XQ, Xu YY, Pen QL, Wang B, Zhu YQ, Tian Y. The incidence and risk factors of related lymphedema for breast cancer survivors post-operation: a 2-year follow-up prospective cohort study. Breast Cancer. 2018 May;25(3):309-314. doi: 10.1007/s12282-018-0830-3. Epub 2018 Feb 3. PMID 29397555
- [Background] Yusof KM, Avery-Kiejda KA, Ahmad Suhaimi S, Ahmad Zamri N, Rusli MEF, Mahmud R, Saini SM, Abdul Wahhab Ibraheem S, Abdullah M, Rosli R. Assessment of Potential Risk Factors and Skin Ultrasound Presentation Associated with Breast Cancer-Related Lymphedema in Long-Term Breast Cancer Survivors. Diagnostics (Basel). 2021 Jul 21;11(8):1303. doi: 10.3390/diagnostics11081303. PMID 34441238
- [Background] Yakut, Y., Yurt, Y., Yağci, G., & Şimşek, İ. E. (2021). Quebec Yardımcı Teknoloji Kullanıcı Memnuniyeti Değerlendirme 2.0 Anketi'nin protez ve ortez kullanan bireylerde Türkçe adaptasyonu. Journal of Exercise Therapy and Rehabilitation, 7(3), 284-295. https://dergipark.org.tr/en/pub/jetr/issue/59488/706401
- [Background] Turna, I. F. (2020). Lenfödem Tanı ve Tedavisine Güncel Bakış. Acibadem Universitesi Saglik Bilimleri Dergisi, 11(1), 0-0. https://doi.org/10.31067/0.2020.238
- [Background] Tidhar D, Armer JM, Deutscher D, Shyu CR, Azuri J, Madsen R. Measurement Issues in Anthropometric Measures of Limb Volume Change in Persons at Risk for and Living with Lymphedema: A Reliability Study. J Pers Med. 2015 Sep 30;5(4):341-53. doi: 10.3390/jpm5040341. PMID 26437431
- [Background] Taghian NR, Miller CL, Jammallo LS, O'Toole J, Skolny MN. Lymphedema following breast cancer treatment and impact on quality of life: a review. Crit Rev Oncol Hematol. 2014 Dec;92(3):227-34. doi: 10.1016/j.critrevonc.2014.06.004. Epub 2014 Jul 2. PMID 25085806
- [Background] Sun F, Hall A, Tighe MP, Brunelle CL, Sayegh HE, Gillespie TC, Daniell KM, Taghian AG. Perometry versus simulated circumferential tape measurement for the detection of breast cancer-related lymphedema. Breast Cancer Res Treat. 2018 Nov;172(1):83-91. doi: 10.1007/s10549-018-4902-z. Epub 2018 Jul 30. PMID 30062571
- [Background] Shi B, Lin Z, Shi X, Guo P, Wang W, Qi X, Zhou C, Zhang H, Liu X, Iv A. Effects of a lymphedema prevention program based on the theory of knowledge-attitude-practice on postoperative breast cancer patients: A randomized clinical trial. Cancer Med. 2023 Jul;12(14):15468-15481. doi: 10.1002/cam4.6171. Epub 2023 Jun 17. PMID 37329176
- [Background] Pappalardo M, Starnoni M, Franceschini G, Baccarani A, De Santis G. Breast Cancer-Related Lymphedema: Recent Updates on Diagnosis, Severity and Available Treatments. J Pers Med. 2021 May 12;11(5):402. doi: 10.3390/jpm11050402. PMID 34065795
- [Background] Ostby PL, Armer JM, Smith K, Stewart BR. Patient Perceptions of Barriers to Self-Management of Breast Cancer-Related Lymphedema. West J Nurs Res. 2018 Dec;40(12):1800-1817. doi: 10.1177/0193945917744351. Epub 2017 Nov 30. PMID 29191123
- [Background] Ostby PL, Armer JM, Dale PS, Van Loo MJ, Wilbanks CL, Stewart BR. Surveillance recommendations in reducing risk of and optimally managing breast cancer-related lymphedema. J Pers Med. 2014 Aug 18;4(3):424-47. doi: 10.3390/jpm4030424. PMID 25563360
- [Background] Sheikhi-Mobarakeh Z, Yarmohammadi H, Mokhatri-Hesari P, Fahimi S, Montazeri A, Heydarirad G. Herbs as old potential treatments for lymphedema management: A systematic review. Complement Ther Med. 2020 Dec;55:102615. doi: 10.1016/j.ctim.2020.102615. Epub 2020 Nov 9. PMID 33221590
- [Background] McLaughlin SA, Brunelle CL, Taghian A. Breast Cancer-Related Lymphedema: Risk Factors, Screening, Management, and the Impact of Locoregional Treatment. J Clin Oncol. 2020 Jul 10;38(20):2341-2350. doi: 10.1200/JCO.19.02896. Epub 2020 May 22. No abstract available. PMID 32442064
- [Background] Li MM, Wu PP, Qiang WM, Li JQ, Zhu MY, Yang XL, Wang Y. Development and validation of a risk prediction model for breast cancer-related lymphedema in postoperative patients with breast cancer. Eur J Oncol Nurs. 2023 Apr;63:102258. doi: 10.1016/j.ejon.2022.102258. Epub 2022 Dec 31. PMID 36821887
- [Background] Kayiran O, De La Cruz C, Tane K, Soran A. Lymphedema: From diagnosis to treatment. Turk J Surg. 2017 Jun 1;33(2):51-57. doi: 10.5152/turkjsurg.2017.3870. eCollection 2017. PMID 28740950
- [Background] Harrington S, Gilchrist L, Sander A. Breast Cancer EDGE Task Force Outcomes: Clinical Measures of Pain. Rehabil Oncol. 2014;32(1):13-21. PMID 25346950
- [Background] Hameeteman M, Verhulst AC, Vreeken RD, Maal TJ, Ulrich DJ. 3D stereophotogrammetry in upper-extremity lymphedema: An accurate diagnostic method. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):241-7. doi: 10.1016/j.bjps.2015.10.011. Epub 2015 Oct 22. PMID 26590631
- [Background] Gandhi A, Xu T, DeSnyder SM, Smith GL, Lin R, Barcenas CH, Stauder MC, Hoffman KE, Strom EA, Ferguson S, Smith BD, Woodward WA, Perkins GH, Mitchell MP, Garner D, Goodman CR, Aldrich M, Travis M, Lilly S, Bedrosian I, Shaitelman SF. Prospective, early longitudinal assessment of lymphedema-related quality of life among patients with locally advanced breast cancer: The foundation for building a patient-centered screening program. Breast. 2023 Apr;68:205-215. doi: 10.1016/j.breast.2023.02.011. Epub 2023 Feb 24. PMID 36863241
- [Background] Fajdic J, Djurovic D, Gotovac N, Hrgovic Z. Criteria and procedures for breast conserving surgery. Acta Inform Med. 2013 Mar;21(1):16-9. doi: 10.5455/AIM.2013.21.16-19. PMID 23572855
- [Background] Donahue PMC, MacKenzie A, Filipovic A, Koelmeyer L. Advances in the prevention and treatment of breast cancer-related lymphedema. Breast Cancer Res Treat. 2023 Jul;200(1):1-14. doi: 10.1007/s10549-023-06947-7. Epub 2023 Apr 27. PMID 37103598
- [Background] Cau N, Galli M, Cimolin V, Grossi A, Battarin I, Puleo G, Balzarini A, Caraceni A. Quantitative comparison between the laser scanner three-dimensional method and the circumferential method for evaluation of arm volume in patients with lymphedema. J Vasc Surg Venous Lymphat Disord. 2018 Jan;6(1):96-103. doi: 10.1016/j.jvsv.2017.08.014. PMID 29248110
- [Background] Boyages J, Xu Y, Kalfa S, Koelmeyer L, Parkinson B, Mackie H, Viveros H, Gollan P, Taksa L. Financial cost of lymphedema borne by women with breast cancer. Psychooncology. 2017 Jun;26(6):849-855. doi: 10.1002/pon.4239. Epub 2016 Aug 21. PMID 27479170
- [Background] Armer JM, Hulett JM, Bernas M, Ostby P, Stewart BR, Cormier JN. Best Practice Guidelines in Assessment, Risk Reduction, Management, and Surveillance for Post-Breast Cancer Lymphedema. Curr Breast Cancer Rep. 2013 Jun;5(2):134-144. doi: 10.1007/s12609-013-0105-0. PMID 26246870
- [Background] Ozhanli Y, Akyolcu N. Satisfaction of Patients with Triage and Nursing Practice in Emergency Departments. Florence Nightingale J Nurs. 2020 Mar 6;28(1):49-60. doi: 10.5152/FNJN.2020.18041. eCollection 2020 Feb. PMID 34263185